CLINICAL TRIAL: NCT03890276
Title: Field Validation of Training Materials and Methods to Build Capacity of Skilled Birth Attendants at Labor and Birth in the Helping Mothers Survive Module 'Essential Care for Labor & Birth' to Improve Quality of Care in Zanzibar
Brief Title: Field Study of Health Worker Training on Helping Mothers Survive Module 'Essential Care for Labor & Birth' in Zanzibar
Acronym: HMS-ECL&B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jhpiego (Other)
Collaborators: Laerdal Foundation (Other); Ministry of Health and Social Welfare, Zanzibar (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB9400
Record Dates: First submitted 2019-03-20; First posted 2019-03-26 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Parturition
Keywords: labor; birth; routine care; midwifery; Zanzibar; Sub-Saharan Africa; training; skilled birth attendant; competency; simulation; video

STUDY DESIGN:
Intervention Model Description: This is a quasi-experimental two-arm study that is a formative, pre- and post-training assessment of healthcare providers who receive the training intervention. In the experimental arm, participants (health care providers) will receive training supplemented with videos. In the comparison arm, participants (heath care providers) will receive training with no video. Participants come from 36 health facilities. There are 18 health facilities sending participants, per study arm.
Who Masked: Outcomes Assessor
Masking Description: Jhpiego data analysts will be blinded to which participants were in which arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HMS EL&C training without video (Active Comparator): Participant health care providers will receive a 1-2 day training in the new 'Helping Mothers Survive Essential Labor and Childbirth' (HMS EL&C) training module. They will be able to: 1) distinguish normal and abnormal findings, 2) competently and confidently manage normal labor and birth to help prevent complications, 3) employ evidence-based practices, 4) rapidly identify and manage complications when they arise and 5) provide respectful care
  Interventions: Other: HMS EL&C training module
- HMS training with video supplementation (Experimental): Participant health care providers will receive a 1-2 day training in the new 'Helping Mothers Survive Essential Labor and Childbirth' (HMS EL&C) training module. They will ALSO receive the training with interspersed with short video clips that that aim to improve understanding and skills acquisition ('Videos used to supplement live trainer'). Video supplementation is meant to standardize the cascaded training in the future as the training is offered at a much larger scale in low and middle income countries.
  Interventions: Other: HMS EL&C training module; Other: Videos used to supplement live trainer

INTERVENTIONS:
Other: HMS EL&C training module — No additional information
Other: Videos used to supplement live trainer — [Cherrie to add]
  Arms: HMS training with video supplementation

SUMMARY:
The goal of this study is to ensure that the training materials and methods for the training module Helping Mothers Survive Essential Care for Labor & Birth (ECL&B) are usable and acceptable by trainers and healthcare providers in Zanzibar. Findings from this study will be used to improve the modules and validate the trainee assessments. This study also compares provider learning outcomes in the training module delivered with and without video demonstration.

Focusing on the first two phases of the Kirkpatrick model, the field validation will answer the following research questions:

1. How acceptable and appropriate for adequate teaching and learning is the training module?
2. What is the gain in knowledge, clinical decision-making, communication, and psychomotor skills of the trainees from pre to post-training assessment? (immediate learner outcomes)
3. Is there a difference in immediate learner outcomes in training where video clips are used during training to supplement live trainer demonstration compared to training where video is not used as a supplement?

DETAILED DESCRIPTION:
The goal of this study is to ensure that the training materials and methods for the training module Helping Mothers Survive Essential Care for Labor & Birth (ECL&B) are usable and acceptable by trainers and healthcare providers in Zanzibar prior to implementing the training. Findings from this study will be used to improve the modules and validate the trainee assessments. This study also compares provider learning outcomes in the training module delivered with and without video demonstration.

Focusing on the first two phases of the Kirkpatrick model, the field validation is designed to answer the following research questions:

1. How acceptable and appropriate for adequate teaching and learning is the training module?
2. What is the gain in knowledge, clinical decision-making, communication, and psychomotor skills of the trainees from pre to post-training assessment? (immediate learner outcomes)
3. Is there a difference in immediate learner outcomes in training where video clips are used during training to supplement live trainer demonstration compared to training where video is not used as a supplement?

Background: To improve the quality of antenatal, intrapartum, and postpartum care, and thus reduce maternal and newborn morbidity and mortality, Jhpiego, in conjunction with global partners, has developed Helping Mothers Survive (HMS), a suite of training modules for frontline providers to use in low- and middle-income countries. HMS is a series of one or two-day, hands-on training modules followed by low-dose, high-frequency (LDHF) practice and other quality improvement activities. These modules are delivered at the worksite to provide ongoing support for clinical performance after training.

The importance of high-quality care during routine labor and birth to ensure the survival of women and their newborns cannot be overstated. The third module in the HMS series addresses the training needs for care during normal labor and birth (ECL&B). The ECL&B module is based on latest WHO guidance.

HMS training modules are developed to specifically address this gap with a plan for "low dose, high frequency" training to offer "boosters" to ensure competency in individual clinical areas and to consolidate skills through practice after training. Local health facility-based providers are responsible for leading short, frequent refresher practice sessions with their peers. Trained providers also conduct quality improvement activities and offer initial simulation-based training for new employees. This emphasis on local capacity building within health facilities makes validation of this training method and accompanying materials important. In addition, because this training will ultimately be disseminated at a larger scale, it is vital that the materials and methods be tested in resource-limited settings at this early stage.

As training in the Helping Mothers Survive modules becomes more widely available through a variety of partner organizations, a concern is that local trainers' skills demonstrations will have high variability in terms of the quality of the training demonstrations resulting in variation in acquisition of learner competencies. This study will investigate whether HMS ECL&B training using in-person trainer supplemented with video demonstrations for several key skills results in better learner competencies immediately post-training compared to the same training with live trainers only.

This mixed-methods, quasi-experimental two-arm study is formative and a pre- and post-training assessment of the training intervention. In the experimental arm, participants (clinicians also called skilled birth attendants) will receive training supplemented with video. In the comparison arm, participants will receive training with no video. This study is similar to the field validation studies for the Bleeding After Birth (BAB) module (Johns Hopkins Bloomberg School of Public Health IRB #0004062) and the BAB+ and Pre-eclampsia/Eclampsia (PE&E) modules (IRB #0007038), completed in 2012 and 2016, respectively, with the addition of an evaluation of video use as a supplement to a live trainer using the HMS training materials.

To assess acceptability of the intervention, focus groups with trainers and providers will be conducted. To assess clinicians' learning in the HMS modules and skill acquisition, there will be knowledge tests, a confidence assessment and three objective structured clinical examination scenarios. Participants' characteristics and past clinical experience will be measured through the self-administered survey.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare providers
* Clinically active birth attendants (defined as having attended or assisted with at least 1 birth in the last month or 3 births in the last 3 months)
* Aged 18 years or older
* Working in government health facilities in Zanzibar

Exclusion Criteria:

-Unable to attend the pre-training and post-training assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
The health care provider's ' 'mean percent correct score' on the Objective Structured Clinical Exam (OSCE) | 1 day post-training
  The mean percent of items answered or performed correctly on OSCE, a simulation of offering care

SECONDARY OUTCOMES:
Percentage of providers who score above the passing threshold of 80% correct on OSCE ('pass rate') | 1 day post-training
  Percentage of providers who score above the passing threshold of 80% correct on OSCE

CONTACTS AND LOCATIONS:
Overall Officials: Cherrie Evans, CNM, DrPH, Principal Investigator — Jhpiego
Locations (6):
- Tanzania (6):
  - Makunduchi Hospital, Makunduchi, Zanzibar
  - Chukwani PHCU+, Mbweni, Zanzibar
  - Chakechake Hospital, Pemba, Zanzibar
  - Wete Hospital, Pemba, Zanzibar
  - Fuoni Primary Health Care Unit +, Stone Town, Zanzibar
  - Mnazi Mmoja Hospital, Stone Town, Zanzibar

IPD SHARING:
Plan to Share IPD: Yes
Any indirect identifiers and facility names will be stripped from the datasets. Data on learning on assessment tools may be made available to other researchers with a signed Data Use Agreement.
Supporting Information: ICF
Time Frame: Jan 10, 2020
Access Criteria: Undetermined

REFERENCES:
- [Background] Evans CL, Bazant E, Atukunda I, Williams E, Niermeyer S, Hiner C, Zahn R, Namugerwa R, Mbonye A, Mohan D. Peer-assisted learning after onsite, low-dose, high-frequency training and practice on simulators to prevent and treat postpartum hemorrhage and neonatal asphyxia: A pragmatic trial in 12 districts in Uganda. PLoS One. 2018 Dec 17;13(12):e0207909. doi: 10.1371/journal.pone.0207909. eCollection 2018. PMID 30557350
- [Background] Evans CL, Johnson P, Bazant E, Bhatnagar N, Zgambo J, Khamis AR. Competency-based training "Helping Mothers Survive: Bleeding after Birth" for providers from central and remote facilities in three countries. Int J Gynaecol Obstet. 2014 Sep;126(3):286-90. doi: 10.1016/j.ijgo.2014.02.021. Epub 2014 Apr 24. PMID 24834851
- See also: Journal Article — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0207909